CLINICAL TRIAL: NCT05431296
Title: Glucose Monitoring After Acute Myocardial Infarct in People With Diabetes
Acronym: GLAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21CX7252
Record Dates: First submitted 2022-06-13; First posted 2022-06-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes; Acute Myocardial Infarction; Acute Myocardial Infarction With ST Elevation; Diabetes Complications
MeSH Terms: conditions — Diabetes Mellitus, Type 2; ST Elevation Myocardial Infarction; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Real time CGM post acute myocardial infarct (Experimental): Real time Dexcom ONE CGM system to be applied for 26 weeks post acute myocardial infarct. Option for participants in this group to continue using rCGM in an open label observational extension phase for a total of 3 years.
  Interventions: Device: Dexcom ONE Continuous Glucose Monitoring System
- Blinded CGM post acute myocardial infarct (No Intervention): Blinded Dexcom ONE CGM system to be applied for 10 days at recruitment, and then at days 17-23, week 10 and week 24. This will be for the purposes of monitoring glucose only and is not an intervention and is blinded to the participants and the study investigators. CGM measurements will be blinded until the end of the study. Management of diabetes in this cohort as per usual standards of care.
- Blinded CGM historical acute myocardial infarct (>6 months and <10 years ago) (No Intervention): Blinded Dexcom ONE CGM system to be applied for 10 days at recruitment. This will be for the purposes of monitoring glucose only and is not an intervention and is blinded to the participants and the study investigators. Management of diabetes in this cohort as per usual standards of care.
- Cardiovascular outcomes control group (No Intervention): Age and sex-matched controls from the NIHR Cardiovascular Health Informatics Collaborative.

INTERVENTIONS:
Device: Dexcom ONE Continuous Glucose Monitoring System — The Dexcom ONE is comprised of a sensor, transmitter and display device (receiver and/or compatible smart device). The system features a redesigned, one-touch auto-applicator and sleek, discreet transmitter. CGM involves insertion of a small plastic cannula to the subcutaneous tissue of the abdominal skin by members of the study team. The cannula is attached to a small data. The cannula is attached to a small transmitter which is taped to the skin and sends data about interstitial glucose via Bluetooth to a receiver which displays a blood glucose reading. The Dexcom G6 sends glucose readings to a compatible smart device or the Dexcom receiver every 5 minutes.
  Arms: Real time CGM post acute myocardial infarct

SUMMARY:
Glucose monitoring after Acute Myocardial infarct in people with diabetes is a Dexcom funded study that is investigating whether the use of continuous glucose monitors (Dexcom ONE model) in people with type 2 diabetes facilitates time in glycaemic range in the 6 months after an acute myocardial infarction. As an exploratory outcome it will investigate whether time in glycaemic range is associated with changes in mortality and major adverse cardiac events in the 6 months after acute myocardial infarct.

DETAILED DESCRIPTION:
The study

1. Patients recruited from cardiology services after ACS (n=140 participants)

   Following informed consent study participants with known diabetes who have had an acute myocardial infarct will be recruited. Participants will be randomly allocated to either the intervention group, referred to as cohort 'a', or to the control group, referred to cohort 'b'. They will be randomised using permuted blocks in a 5:2 ratio (intervention:control). CGM (real-time or blinded) will be applied to participants prior to discharge.

   Following hospital discharge, the effects of changes in blood glucose levels on cardiac and health outcomes will be evaluated. Participants recruited to cohort 'a' will wear real-time CGM continuously after hospital discharge for 26 weeks. They will have face-to-face, telephone or video reviews of CGM data at 4 and 12 weeks with clinician-led diabetes treatment escalation according to NICE guidelines based aiming for >70% time in target blood glucose range, 3.9-10mmol/L (50% for older or high risk individuals). Participants recruited to cohort 'b' will wear blinded CGM for 10 days after insertion. They will wear blinded CGM again for 10 days , with the second sensor insertion at days 17-23, third sensor insertion during week 10 and fourth sensor insertion during week 24. Following each sensor wear, participants in cohort 'b' will have a study visit when their sensor data will be downloaded. Participants in cohort 'b' will receive face-to-face or remote support to insert and establish blinded CGM but no clinical review and the participant should manage their diabetes as the participant normally would. At 26 weeks data will be analysed for all primary and secondary outcomes.

   The participants who receive real-time CGM will be compared to age and sex-matched controls, who's data will be obtained from the NIHR Cardiovascular Health Informatics Collaborative for comparison of cardiovascular outcomes.

   At 26 weeks data (clinical details of hospital admissions, further cardiac events, medication changes, blood test results obtained from hospital records and on discussion with the participant) will be collected for all primary and secondary outcomes. Imperial College Healthcare NHS Trust uses an electronic patient record system that is connected to the central NHS Spine and is updated in real-time. People who have died, even if the person has died out of hospital, will be recorded as deceased and this will be visible to the research team. End of study will be defined as Last Subject Last Visit (LSLV) at which point the participant will be asked to return or post back their study equipment and the participant will revert to standard care with their usual GP, community or hospital diabetes team.

   If participants in cohort 'a' wish to continue real time CGM beyond the primary endpoint, they will be given the opportunity to continue to use CGM in an open label observation phase for three years from the start of the study. The study will continue to supply all CGM equipment to participants. The participant's GP, and if appropriate, specialist diabetes team, will be made aware that they are continuing on CGM for research purposes. The CGM data will continue to be collected by the study team for research purposes and the participant will have 6 monthly contact from the study team by telephone, virtually, in person or by email, in line with the participant's preference. The purpose of these visits will be to give CGM supplies, check that the participant still wishes to continue on CGM, and to gather information on diabetes medications, and major adverse cardiac events.

   The study team will not be managing the participant's diabetes over the extension phase and their diabetes care will revert to the team who had previously managed it. During the observational phase, the trial team will not directly make changes to diabetes care on the basis of the results of the additional CGM but results that are significant to the participant's care, or any incidental findings, will be transmitted to their usual care giver and this may result in changes to their diabetes management. It is not anticipated that there will be incidental findings. Participants will be encouraged to contact the study team if they have any problems or concerns in relation to the ongoing use of the sensors.

   Eligible participants admitted to the Hammersmith Hospital HAC with confirmed ACS will be recruited as soon as possible after hospital admission. Patients lacking capacity to consent will not be recruited. During admission, HbA1c levels will be sent as part of routine blood testing.

   The research team will collect full medical and medication history, as well as historic bloods test results from the hospital computer systems as per routine clinical care. All participants recruited during their hospital admission will have blood tests (for HbA1c and other markers of metabolism) during admission and at 4, 12 and 24-26 weeks.

   Participants in cohorts 'a' and 'b' will be asked to complete the Diabetes Treatment Satisfaction Scale questionnaire, the Audit of Diabetes Dependent Quality of Life questionnaire and the Hypoglycaemia Symptom Rating Questionnaire at the time of recruitment, and then at 4, 12, and 24 weeks. Participants will also be asked to fill out an Audit of Diabetes Dependent Quality of Life-19 questionnaire at the time of recruitment and at 12 and 24 weeks.
2. Patients recruited from diabetes and cardiology clinics after ACS (n=20 participants)

   Eligible participants reviewed in clinic with confirmed previous ACS will be recruited. Patients lacking capacity to consent will not be recruited. HbA1c levels will be sent as part of routine blood testing. The research team will collect full medical and medication history, as well as historic bloods test results from the hospital computer systems as per routine clinical care.

   Blinded CGM will be applied to 20 participants with a history of ACS more than 6 months ago, but less than 10 years ago and a known diagnosis of type 2 diabetes who take one or oral diabetic agents, and/or GLP 1 receptor analogue, and/or insulin. The blinded CGM will be worn for 10 days and then returned to (or collected by) the study team.

   These participants be asked to complete a Diabetes Treatment Satisfaction Scale questionnaire, the Audit of Diabetes Dependent Quality of Life questionnaire and the Hypoglycaemia Symptom Rating Questionnaire at the time of recruitment. The participants will have a blood test looking at glycaemic control and markers of metabolism at the time of recruitment.
3. Data collection from the Health Information Collaborative

The participants who receive real-time CGM will be compared to age and sex-matched controls, who's data will be obtained from the NIHR Cardiovascular Health Informatics Collaborative for comparison of cardiovascular outcomes. Imperial College Healthcare NHS Trust has led the NIHR Cardiovascular Health Informatics Collaborative, which was established to enable the sharing and repurposing of routinely captured clinical data for re-use in research. Clinical patient data is extracted and put into a tabular format which includes demographics, emergency department attendance, inpatient episodes, blood tests, diagnoses, operations and procedures, echocardiography measurements and survival status. This infrastructure has been used to investigate patient outcomes in previous studies and will provide endpoint data for the patients enrolled into this study.

2. Clinical study recruitment: Single Centre- Imperial College Healthcare NHS Trust Design: Randomised control trial

Population:

Interventional cohort: 100 participants with type 2 diabetes and acute myocardial infarction will wear real time CGM for 26 weeks Control: 40 participants with type 2 diabetes and acute myocardial infarction will wear blinded CGM for 10 days at 4 time points in the 6 months after infarct.

Clinic cohort: 20 participants with type 2 diabetes who have had a myocardial infarct > 6 months ago but <10 years ago will wear blinded CGM for 10 days.

Case control: NIHR Cardiovascular Health Informatics Collaborative dataset

Timescale: Each participant will be in the trial for 6 months. It is anticipated that it will take 18-24 months to recruit to target study number.

3. Statistics The study is powered to detect a change of between 7.2 and 13.2% difference in time in range glucose 3.9-10mmol/l between the real time and blinded CGM groups at 6 months depending the standard deviation used in the power calculation with two tailed alpha of 0.05 and power of 80%. This difference is thought to be a clinically meaningful and achievable difference.

For each questionnaire, mean ± SD values or percentiles appropriate to the distribution will be given by randomization group for the total score and each subscale. Treatment group comparisons will be made using linear models.

The following tabulations will be performed according to treatment group without statistical testing: baseline demographics and clinical characteristics, protocol deviations, device malfunctions and other reported device issue.

For all CGM outcomes, a multilevel model of repeated measures (MMRM) will be used.

4. Data During the course of the study visits some data will be stored on laptop computers, not connected to the Internet, for later statistical analysis. These data will be coded and non- identifiable. Laptop computers may be used during the visits for portability and convenience. At the end of each visit the anonymised data will be transferred immediately to a secure web-server (details below) and will be deleted from the laptop.

Any identifiable participant data will be stored in a locked filing cabinet in a secure room in each investigation centre. Only clinical research team will have access to this participant identifiable data.

5. Adverse Events (AEs) Reporting Procedures. All adverse events will be reported. Depending on the nature of the event the reporting procedures below will be followed. Any questions concerning adverse event reporting will be directed to the Chief Investigator in the first instance.

Non serious AEs: All such events will be recorded. Serious Adverse Events (SAEs): An SAE form will be completed and faxed to the Chief Investigator within 24 hours. However, hospitalisations for elective treatment of a pre-existing condition do not need reporting as SAEs.

Reports of related and unexpected SAEs will be submitted within 15 days of the Chief Investigator becoming aware of the event. The Chief Investigator will also notify the Sponsor of all SAEs, where in the opinion of the Chief Investigator, the event is:

'related', i.e. resulted from the administration of any of the research procedures; and 'unexpected', i.e. an event that is not listed in the protocol as an expected occurrence Local investigators will report any SAEs as required by their Local Research Ethics Committee, Sponsor and/or Research & Development Office.

ELIGIBILITY:
Inclusion Criteria:

From the Hammersmith Hospital In-patient Cardiology Services:

* Adults aged >18 years
* Known or newly diagnosed type 2 diabetes
* Taking one or more oral hypoglycaemic agent, GLP1 receptor analogue and/or insulin
* Admitted to Hammersmith Hospital cardiology inpatient services with ACS
* Raised blood troponin level on admission

From Imperial College Healthcare Trust Diabetes and Cardiology Clinics:

* Adults aged >18 years
* Known type 2 diabetes
* Previous acute coronary syndrome within the last 10 years but > 6 months ago
* Taking one or more oral hypoglycaemic agent and /or GLP1 receptor analogue, and/or insulin

Exclusion Criteria:

From the Hammersmith Hospital In-patient Cardiology Services:

* HbA1c <48mmol/mol
* People who have previously had bariatric surgery
* People taking hydroxyurea
* People who undergo haemodialysis or peritoneal dialysis
* Unable to participate due to other factors, as assessed by the Chief Investigators
* Pregnancy as determined by clinical team
* Known to have a terminal condition or conditions that suggest a life expectancy less than 1 year

From Imperial College Healthcare Trust Diabetes and Cardiology Clinics:

* HbA1c <48mmol/mol
* People who have previously had bariatric surgery
* People taking hydroxyurea
* People who undergo haemodialysis or peritoneal dialysis
* Unable to participate due to other factors, as assessed by the Chief Investigators
* Pregnancy as determined by clinical team
* Known to have a terminal condition or conditions that suggest a life expectancy less than 1 year
* Previous acute coronary syndrome more than 10 years ago or within the last 6 months

Withdrawal criteria

* The subject has a serious event related to the study
* Investigated initiated discontinuation of study due to participation or equipment concerns
* Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Percent time spent in glucose target range (3.9-10mmol/L) | 26 weeks
  Percent time spent in glucose target range (3.9-10mmol/L)

SECONDARY OUTCOMES:
Number hypoglycaemic excursions. | 26 weeks
  Number of detected excursions on CGM to glucose <3.9mmol/L
Time spent in hypoglycaemia (<3.9mmol/L, 70mg/dL; <3.0mmol/L, 54mg/dL), | 26 weeks
  Time spent with glucose <3.9mmol/L, time spent with glucose <3mmol/L
Time in euglycaemia (3.9-7.8mmol/L, 70-140mg/dL). | 26 weeks
  Secondary outcome
Time in hyperglycaemia (>10mmol/L, 180mg/dL). | 26 weeks
  Secondary outcome
Hypoglycaemia requiring 3rd party assistance. | 26 weeks
  Number of hypoglycaemia events requiring assistance of 3rd party
Number hypoglycaemic excursions (sensor glucose <3.0mmol/l for >= 20min) | 26 weeks
  Secondary outcome
HbA1c at 12 weeks and 26 weeks. | 26 weeks
  Glycosylated haemoglobin (HbA1c) in percent or mmol/mol
Glucose variability assessed by %Coefficient of Variation (%CV). | 26 weeks
  Variability of glucose (oscillations in glucose values)
Mean Absolute Glucose (MAG) | 26 weeks
  mean absolute Mean absolute glucose change per unit time
Health and treatment-related quality of life measured by the Diabetes Treatment Satisfaction Scale score. | 26 weeks
  The DTSQ s (status version) and DTSQ c (change version) contain eight items each, six of them (questions 1 and 4-8) measure the Treatment Satisfaction and questions 2 and 3, concerning Perceived Frequency of Hyperglycaemia ('Perceived Hyperglycaemia')/Perceived Frequency of Hypoglycaemia ('Perceived Hypoglycaemia') respectively, are treated separately from the satisfaction items and from each other. DTSQs scores range from 6 = very satisfied to 0 = very dissatisfied and DTSQc scores from +3 = much more satisfied now to -3 = much less satisfied now, with 0 (midpoint), representing no change.
Hypoglycaemic symptoms | 26 weeks.
  The HypoSRQ is designed to measure the experience of common symptoms associated with hypoglycaemia in people with diabetes. This questionnaire has 18 questions- which require a yes/no response. If the answer is yes, the participant then grades the symptom against 4 categories of severity
Low Blood Glucose Index (LBGI}) | 26 weeks.
  Secondary Outcome
Audit of Diabetes Dependent Quality of Life questionnaire domain. | 26 weeks.
  The Audit of Diabetes Dependent Quality of Life -19 questionnaire is a 19 item measure that looks at the impact of diabetes on specific aspects of life and the importance of these aspects for QoL.

OTHER OUTCOMES:
MACE endpoint defined as death due to cardiac cause or hospitalisation with acute coronary syndrome (including MI and unstable angina); heart failure; unscheduled revascularisation; arrhythmia; cerebrovascular event | 26 weeks
  Exploratory outcome
All cause mortality | 26 weeks
  Exploratory outcome
Duration of hospital admission before 'medically fit for discharge'. | 26 weeks
  Exploratory outcome
Escalation to High Dependency Unit or Intensive Care Unit during primary hospital episode. | 26 weeks
  Exploratory outcome
Echocardiographic measurements of cardiac function. | 26 weeks
  Ejection fraction as a percentage
Changes in care, measured by changes in diabetes medication usage. | 26 weeks
  Exploratory outcome

CONTACTS AND LOCATIONS:
Overall Officials: Monika Reddy, MBChB, PhD, Principal Investigator — Imperial College London; Jamil Mayet, MBChB, MD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital inpatient cardiology services, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malmberg K, Ryden L, Hamsten A, Herlitz J, Waldenstrom A, Wedel H. Mortality prediction in diabetic patients with myocardial infarction: experiences from the DIGAMI study. Cardiovasc Res. 1997 Apr;34(1):248-53. doi: 10.1016/s0008-6363(96)00263-5. PMID 9217897
- [Background] Cheung NW, Wong VW, McLean M. The Hyperglycemia: Intensive Insulin Infusion in Infarction (HI-5) study: a randomized controlled trial of insulin infusion therapy for myocardial infarction. Diabetes Care. 2006 Apr;29(4):765-70. doi: 10.2337/diacare.29.04.06.dc05-1894. PMID 16567812
- [Background] Malmberg K, Ryden L, Efendic S, Herlitz J, Nicol P, Waldenstrom A, Wedel H, Welin L. Randomized trial of insulin-glucose infusion followed by subcutaneous insulin treatment in diabetic patients with acute myocardial infarction (DIGAMI study): effects on mortality at 1 year. J Am Coll Cardiol. 1995 Jul;26(1):57-65. doi: 10.1016/0735-1097(95)00126-k. PMID 7797776
- [Background] Jackson MA, Ahmann A, Shah VN. Type 2 Diabetes and the Use of Real-Time Continuous Glucose Monitoring. Diabetes Technol Ther. 2021 Mar;23(S1):S27-S34. doi: 10.1089/dia.2021.0007. PMID 33534631
- [Background] Karter AJ, Parker MM, Moffet HH, Gilliam LK, Dlott R. Association of Real-time Continuous Glucose Monitoring With Glycemic Control and Acute Metabolic Events Among Patients With Insulin-Treated Diabetes. JAMA. 2021 Jun 8;325(22):2273-2284. doi: 10.1001/jama.2021.6530. PMID 34077502
- [Background] Yapanis M, James S, Craig ME, O'Neal D, Ekinci EI. Complications of Diabetes and Metrics of Glycemic Management Derived From Continuous Glucose Monitoring. J Clin Endocrinol Metab. 2022 May 17;107(6):e2221-e2236. doi: 10.1210/clinem/dgac034. PMID 35094087
- [Background] Li M, Chen G, Feng Y, He X. Stress Induced Hyperglycemia in the Context of Acute Coronary Syndrome: Definitions, Interventions, and Underlying Mechanisms. Front Cardiovasc Med. 2021 May 12;8:676892. doi: 10.3389/fcvm.2021.676892. eCollection 2021. PMID 34055942
- [Background] Lee W, Kim SH, Yoon CH, Suh JW, Cho YS, Youn TJ, Chae IH. Impact of Long-term Glycosylated Hemoglobin in Patients with Acute Myocardial Infarction: a retrospective cohort study. Sci Rep. 2020 Apr 21;10(1):6726. doi: 10.1038/s41598-020-63802-1. PMID 32317703
- [Background] Lu J, Wang C, Shen Y, Chen L, Zhang L, Cai J, Lu W, Zhu W, Hu G, Xia T, Zhou J. Time in Range in Relation to All-Cause and Cardiovascular Mortality in Patients With Type 2 Diabetes: A Prospective Cohort Study. Diabetes Care. 2021 Feb;44(2):549-555. doi: 10.2337/dc20-1862. Epub 2020 Oct 23. PMID 33097560
- [Background] Bauters C, Lemesle G, de Groote P, Lamblin N. A systematic review and meta-regression of temporal trends in the excess mortality associated with diabetes mellitus after myocardial infarction. Int J Cardiol. 2016 Aug 15;217:109-21. doi: 10.1016/j.ijcard.2016.04.182. Epub 2016 May 4. PMID 27179900
- [Background] Oser TK, Litchman ML, Allen NA, Kwan BM, Fisher L, Jortberg BT, Polonsky WH, Oser SM. Personal Continuous Glucose Monitoring Use Among Adults with Type 2 Diabetes: Clinical Efficacy and Economic Impacts. Curr Diab Rep. 2021 Dec 9;21(11):49. doi: 10.1007/s11892-021-01408-1. PMID 34882273